CLINICAL TRIAL: NCT04028167
Title: Phase II Study of Induction FLOT Followed by Neoadjuvant Chemoradiation in Patients With Resectable Adenocarcinoma of the Esophagus or Gastroesophageal Junction
Brief Title: Induction FLOT With CROSS CRT for Esophageal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Cancer Society, Inc. (Other); Cancer League of Colorado (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0376.cc; P30CA046934 (NIH)
Record Dates: First submitted 2019-06-04; First posted 2019-07-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Adenocarcinoma Esophagus; Adenocarcinoma of the Gastroesophageal Junction
Keywords: Resectable
MeSH Terms: conditions — Adenocarcinoma Of Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sequential FLOT followed by chemoradiation (Experimental): Sequential Chemotherapy with Docetaxel, Oxaliplatin, and 5-Fluorouracil/Leucovorin followed by chemoradiation with concurrent carboplatin and paclitaxel
  Interventions: Drug: Sequential FLOT followed by chemoradiation

INTERVENTIONS:
Drug: Sequential FLOT followed by chemoradiation — Chemotherapy with Docetaxel, Oxaliplatin, and 5-Fluorouracil/ Leucovorin

SUMMARY:
This study evaluates a novel regimen of induction chemotherapy using a combination of docetaxel, oxaliplatin, and leucovorin, with short term infusional 5-FU (FLOT), given prior to chemoradiotherapy with concurrent carboplatin and paclitaxel, as neoadjuvant therapy prior to definitive surgical resection for patients with adenocarcinoma of the esophagus or gastroesophageal junction

DETAILED DESCRIPTION:
Clinical outcomes following standard of care therapy for resectable esophageal and gastroesophageal junction adenocarcinoma are suboptimal, with low rates of pathologic complete response (pCR) to current neoadjuvant treatment strategies. Although significant progress has been made by incorporation of neoadjuvant chemoradiation or perioperative chemotherapy, most patients will ultimately develop disease recurrence, with both locoregional and distant recurrence representing a significant component of failure. For patients receiving preoperative chemoradiation, a regimen consisting of concurrent carboplatin and paclitaxel with radiotherapy has been established as a standard of care based on the Chemoradiotherapy for Esophageal Cancer Followed by Surgery Study (CROSS). In the long term results of CROSS, locoregional progression was noted in 22% of patients receiving neoadjuvant therapy, with distant progression in 39%.

Recent studies have also suggested perioperative chemotherapy as a potential alternative strategy for selected patients, based on results of the MAGIC trial, which included a subset patients with esophageal/GE junction tumor location, and demonstrated improved survival for patients receiving perioperative epirubicin, cisplatin, and infusional 5-fluorouracil (ECF) compared to surgery alone. The FLOT4-AIO trial has subsequently demonstrated a further overall survival benefit to a perioperative regimen of docetaxel, oxaliplatin, and leucovorin, with short term infusional 5-FU (FLOT) compared to ECF. A regimen of perioperative FLOT is currently being compared to preoperative chemoradiotherapy using the CROSS regimen in the ongoing ESOPEC trial (NCT02509286).

Given the significant risk of recurrence either with the CROSS preoperative chemoradiation regimen, or the perioperative FLOT regimen, it is plausible that selected patients may benefit from a combination of intensified systemic therapy using the FLOT backbone, in combination with sequential preoperative chemoradiation due to the known risk of locoregional recurrence in this population. This study evaluates the proposed neoadjuvant regimen of induction FLOT followed by neoadjuvant chemoradiation in patients with resectable cT3/T4 or node positive adenocarcinoma of the esophagus or gastroesophageal junction.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be a male or female aged 18-100.
4. Have newly diagnosed, resectable cT3-T4 or node positive adenocarcinoma of the esophagus or gastroesophageal junction as assessed by CT or MRI of the chest, abdomen and pelvis and by endoscopic ultrasound, with pathologic diagnosis obtained within 3 months of signing consent, without delivery of prior chemotherapy or radiation therapy.
5. Subjects must be previously untreated with systemic chemotherapy or radiation therapy.
6. Subjects must be deemed a candidate for trimodality therapy (radiation, chemotherapy and surgery) based upon multidisciplinary evaluation with plan for preoperative chemoradiation followed by surgical resection.
7. ECOG performance status score of 0-1 (See Appendix).
8. Adequate bone marrow function (WBC > 3 x 109/L; hemoglobin > 9 g/dl; platelets > 100 x 109/L)
9. Adequate liver function (total bilirubin < 1.5 x upper limit of normal, AST < 3 x upper limit of normal, and ALT < 3 x upper limit of normal)
10. Serum creatinine < 1.5 x ULN or calculated creatinine clearance > 50 mL/min (using the Cockcroft-Gault formula)

    Males:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

    Females:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
11. Women of child-bearing potential (WOCBP) must have a negative serum or urine pregnancy test within 2 weeks prior to study enrollment and must agree to follow instructions for method(s) of contraception for the duration of the study period and at least 3 months after the last dose of chemotherapy is administered. For the purpose of this study, a woman is considered of childbearing potential following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

    For the purpose of this study, methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods and acceptable contraception. Such methods include:
    * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:
    * oral
    * intravaginal
    * transdermal
    * progestogen-only hormonal contraception associated with inhibition of ovulation:
    * oral
    * injectable
    * implantable
    * intrauterine device (IUD)
    * intrauterine hormone-releasing system (IUS)
    * bilateral tubal ligation
    * vasectomized partner
    * sexual abstinence
12. WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements but still must undergo pregnancy testing as described in this section.
13. Males who are sexually active with WOCBP must agree to follow instructions for methods of contraception for the duration of the study period and for at least 3 months (duration of sperm turnover) after the last dose of chemotherapy is administered. In addition, males must be willing to refrain from sperm donation during this time.

Azoospermic males are exempt from contraceptive requirements.

Exclusion Criteria:

1. Subjects with metastatic or inoperable esophageal or gastroesophageal junction adenocarcinoma.
2. Subjects with esophageal or gastroesophageal junction squamous cell carcinoma or adenosquamous carcinoma.
3. Prior treatment with chemotherapy or radiation therapy for esophageal or gastroesophageal adenocarcinoma.
4. Prior malignancy active within the previous 3 years that is felt to exclude the patient from definitive therapy of esophageal or gastroesophageal cancer, or if prior cancer therapy is felt by the investigator to significantly increase toxicity risk from the study regimen.
5. Prior history of thoracic or abdominal radiotherapy that would overlap with the planned treatment volume.
6. Active collagen vascular disease.
7. Subjects with > Grade 1 peripheral neuropathy.
8. Any serious or uncontrolled medical disorder or active infection, that in the opinion of the investigator may increase the risk associated with study participation, study treatment administration or would impair the ability of the subject to receive study treatment.
9. Known history of hepatitis B or hepatitis C.
10. Clinically unstable cardiac disease including unstable angina, congestive heart failure, ventricular arrhythmia or known prior QTc > 450msec.
11. History of allergy or hypersensitivity to any of the study drugs or study drug components.
12. Any contraindications to any of the study drugs of the chemotherapy regimens (FLOT or carboplatin/paclitaxel) selected by the investigator. Investigators should refer to the local package insert of the chemotherapy drugs.
13. Prisoners or subjects who are involuntarily incarcerated.
14. History of psychiatric illness that precludes completion of informed consent process, or which is deemed by the investigators as potentially influencing study compliance.
15. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
16. Pregnant or breast-feeding women.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2026-01-02 (Actual); Study Completion 2027-04-19 (Estimated)

PRIMARY OUTCOMES:
Evaluate the rate of pathologic complete response (pCR) to the study regimen. | 5 years
  The percentage of pathologic complete response at resection for patients who has completed the study regimen of induction FLOT, CROSS regimen chemoradiation, and surgical resection

SECONDARY OUTCOMES:
To determine estimates of the 1-year overall survival and disease-free survival among patients treated with the study regimen. | 5 years
  The endpoint of overall survival will be defined by the proportion of evaluable patients that are living at a 1-year time interval from initial pathologic diagnosis. The endpoint of disease-free survival will be defined by the proportion of evaluable patients that are living and free of cancer recurrence at a 1-year time interval from initial pathologic diagnosis
To describe toxicity of the study regimen as a component of neoadjuvant therapy for the study population. | 5 years
  The proportion of patients experiencing any ≥grade 3 and ≥grade 4 toxicity as defined by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be recorded.
Patient reported quality of life | 5 years
  Patient reported quality of life outcomes using the validated European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30)
Measurement of change in the SUVmax on FDG-PET following induction FLOT, compared to initial diagnosis, and describe change in SUVmax among patients with and without a pCR to neoadjuvant therapy. | 5 years
  Percentage reduction in SUVmax from the baseline to the post-chemotherapy PET.
Measurement of ctDNA to generate initial descriptive data regarding ctDNA kinetics as a potential measure of treatment response | 5 years
  The sensitivity and specificity of detectable ctDNA postoperatively to predict 1 year disease-free survival within the study cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Olsen, MD, Principal Investigator — University of Colorado, Denver
Locations (7):
- United States (7):
  - University of Colorado Hospital, Aurora, Colorado
  - UCHealth Southern Colorado - Memorial Hospital Central, Colorado Springs, Colorado
  - UCHealth Southern Colorado - Memorial Hospital North, Colorado Springs, Colorado
  - UCHealth Northern Colorado - Poudre Valley Hospital, Fort Collins, Colorado
  - UCHealth Northern Colorado - Harmony Campus, Fort Collins, Colorado
  - UCHealth Northern Colorado - Greeley Hospital, Greeley, Colorado
  - UCHealth Northern Colorado Medical Center of the Rockies, Loveland, Colorado

IPD SHARING:
Plan to Share IPD: No